CLINICAL TRIAL: NCT04641247
Title: An Open-Label, Multicenter, Long-term Treatment Extension Study in Subjects Who Have Completed a Prior GlaxoSmithKline/TESARO-Sponsored Niraparib Study and Are Judged by the Investigator to Benefit From Continued Treatment With Niraparib
Brief Title: A Long-term Treatment Extension Study of Niraparib in Participants Who Completed a Prior GlaxoSmithKline/TESARO-sponsored Niraparib Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213409; 2020-002667-53 (EudraCT Number); 2023-506618-29 (Registry Identifier: CTIS)
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Neoplasms; Breast Neoplasms
Keywords: Adverse events; Open-label extension; Parent study; Niraparib; Safety
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms | interventions — niraparib

STUDY DESIGN:
Intervention Model Description: Participants will receive niraparib once a day, continuously throughout each 90-day cycle.
Masking Description: This will be an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving niraparib (Experimental): Participants will receive niraparib once a day, continuously throughout each 90-day cycle until one of the following occurs: disease progression, unacceptable toxicity, initiation of new anticancer therapy that was not part of the parent study, withdrawal of consent, discontinuation at the discretion of the Investigator, noncompliance with protocol, death, or discontinuation for any other reason. The doses provided in this long-term treatment extension study will be those defined in the parent study for each enrolled participant. The starting dose of niraparib will be the same as the assigned dose and regimen that were given in the parent study.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib tablets or capsules will be given once a day via the oral route.

SUMMARY:
This is a global extension study to provide continued access to niraparib and further characterize the long-term safety of niraparib treatment in participants who are currently receiving treatment with niraparib within GlaxoSmithKline/TESARO-sponsored studies (NCT01847274, NCT02354586, NCT01905592, NCT03308942, NCT02657889) that has fulfilled the requirements for the primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to understand the study procedures and agrees to participate in the study by providing written informed consent.
* Participant is willing and able to comply with scheduled visits, treatment plans, and any other study procedures.
* Participant is currently receiving treatment with niraparib (as monotherapy or in combination) in a GlaxoSmithKline/TESARO-sponsored study that has fulfilled the requirements for the primary objective.
* Participant is currently benefiting from treatment with niraparib as assessed by the Investigator according to the parent study protocol requirements.
* Participants of childbearing potential who are sexually active and their partners must agree to the use of an effective form of contraception throughout their participation during study treatment through 180 days after last dose of study drug.

Exclusion Criteria:

* Participant has been permanently discontinued from niraparib treatment in the parent study for any reason.
* Participant currently has unresolved toxicities for which niraparib dosing has been interrupted in the parent study. Participants meeting all other eligibility criteria may be enrolled once toxicities have resolved to allow niraparib treatment to resume.
* Participant is pregnant or is expecting to conceive children while receiving study drug or for up to 180 days after the last dose of study drug. Participant is breastfeeding or is expecting to breastfeed within 30 days of receiving the final dose of study drug (women should not breastfeed or store breastmilk for use during niraparib treatment and for 30 days after receiving the final dose of study treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs) and AEs of special interest (AESI) | Up to 5 years
  AEs, SAEs and AESI will be collected.
Number of participants with clinically significant changes in Eastern Co-operative Oncology Group (ECOG) performance status | Up to 5 years
  The performance status will be assessed using ECOG scale, where Grade 0 (fully active), Grade 1 (restricted in physically strenuous activity), Grade 2 (ambulatory and capable of all self-care), Grade 3 (capable of only limited self-care) and Grade 4 (completely disabled). Number of participants with clinically significant changes in ECOG performance status will be summarized.
Number of participants with clinically significant changes in hematology and clinical chemistry parameters | Up to 5 years
  Blood samples will be collected for the analysis of hematology and clinical chemistry parameters.
Number of participants with clinically significant changes in vital signs | Up to 5 years
  Number of participants with clinically significant changes in vital signs will be assessed.
Number of participants with clinically significant changes in physical examination | Up to 5 years
  Number of participants with clinically significant changes in physical examination will be assessed.
Number of participants with use of concomitant medications | Up to 5 years
  Number of participants using concomitant medications will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (13):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Harvey, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
- Austria (2):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Vienna
- Canada (3):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Odense C, Denmark
- France (2):
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
- GSK Investigational Site, Haifa, Israel
- GSK Investigational Site, Cremona, Italy
- GSK Investigational Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.